CLINICAL TRIAL: NCT02577458
Title: Phase 1 Study of the Combination of CM082 With Everolimus in Patients With Metastatic Renal Cell Carcinoma (RCC): Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy
Brief Title: Study of the Combination of CM082 With Everolimus in Patients With mRCC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AnewPharma (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM082-CA-I-103
Record Dates: First submitted 2015-10-12; First posted 2015-10-16 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Renal Cell Carcinoma Recurrent
MeSH Terms: interventions — vorolanib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CM082 plus everolimus (Experimental): CM082 plus everolimus
  Interventions: Drug: CM082; Drug: Everolimus

INTERVENTIONS:
Drug: CM082 — CM082 tablets taken orally once a day on 28-day cycles
  Other Names: X-82
Drug: Everolimus — Everolimus tablets taken orally once a day on 28-day cycles
  Other Names: Affinitor

SUMMARY:
This is a Phase I Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of CM082 in Combination with Everolimus in Chinese Patients With Advanced Renal Cell Carcinoma.

DETAILED DESCRIPTION:
This is a Phase I Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of CM082 in Combination with Everolimus in Chinese Patients With Renal Cell Carcinoma (RCC). After the maximum tolerated dose (MTD) or the optimal biological dose is identified, an expansion cohort of ~10 advanced renal cell carcinoma patients will be enrolled to further characterize the safety and tumor response by CT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of clear cell renal cell carcinoma
* Progressed on at least one standard therapy
* Measurable disease per Recist1.1
* Eastern Cooperative Group (ECOG) Performance Status score of 0 or 1
* Life expectancy of at least 12 weeks
* No abnormal bone marrow function
* Adequate heart, lung, liver, kidney organ system functions, and meet the following requirements:

  * Total bilirubin ≤1.5 times the upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5x the upper limit of normal (ULN) if no liver involvement or ≤5x the upper limit of normal with liver involvement.
  * Creatinine ≤ 1.5 x ULN
  * Urine protein <1+
  * QTcF < 450 ms
  * LVEF ≥ 50%
* At least 4 weeks after receiving cancer therapy (i.e., chemotherapy, radiation therapy, biologic therapy, hormonal therapy); 3 months after surgery and recovered
* Willingness and ability to comply with trial and follow-up procedures
* Ability to understand the nature of this trial and give written informed consent

Exclusion Criteria:

* Currently receiving anti-cancer treatment
* Other tumors in addition to renal cell carcinoma
* Have taken strong cytochrome P450 3A4 inhibitors or inducers in the last 2 weeks
* Concomitant use of drugs with a risk of causing prolonged corrected QT interval and/or Torsades de Pointes
* Patients with a history of intolerance to, or significant toxicity with VEGFR tyrosine kinase inhibitor(s) (TKI) or everolimus
* Females who are pregnant or breastfeeding
* Those in reproductive ages who refuse to use contraception
* Those with concurrent condition(e.g. psychological, neuronal, cardiovascular, respiratory conditions or infections) that in the investigator's opinion would jeopardize compliance with the protocol
* Patients with known central nervous system (CNS) metastases
* Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of CM082 or everolimus
* Patients with known severe lung disorders such as asthma, chronic obstructive pulmonary disease (COPD)
* Patients who are HIV positive
* Drug or alcohol abuser

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-03 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 12 months
  To determine the Maximum Tolerated Dose of the Combination in Chinese RCC Patients

SECONDARY OUTCOMES:
Pharmacokinetics assessed by area under the plasma concentration versus time curve (AUC) of CM082 and everolimus | 12 months
Objective response rate | 18 months
  Objective response rate (ORR)
Progress free survival | 24 months
  Progress free survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, M.D, Study Chair — Peking University Cancer Hospital & Institute; Xinan Sheng, M.D, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China